CLINICAL TRIAL: NCT07181980
Title: Effect of Intercostal Mulligan Moblization on Shoulder Dysfunction Post Mastectomy
Brief Title: Intercostal Mulligan Moblization Post Mastectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Medhat Nagib Abd Elhakim, Submitted In Partial Fulfilment of The Requirements For Master Degree In Department of Physical Therapy for surgery Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005413
Record Dates: First submitted 2025-08-26; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Post Mastectomy Complications
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intercostal mulligan moblization (Active Comparator)
  Interventions: Other: Intercostal mulligan mobilization with shoulder abduction; Other: Exercise
- control group (Active Comparator)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Intercostal mulligan mobilization with shoulder abduction — Intercostal mulligan mobilization with shoulder abduction: is mulligain technique where the patient was Side lying with affected side up and the therapist Therapist placed ulnar side of his hand along the intercostal space of affected rib in oblique direction on the patient's wall of chest. Therapist's other hand hold the patient's elevated arm close to his abdomen 3sets 10 reptations
  * Assistive range of motion exercises (AAROME): Two sets of 15 repetitions of each exercise were performed for AAROME .
  * Active stretching: Two sets of 10 repetitions with 15- sec hold and relax times were performed for active stretching.
  * Strengthening exercises for the shoulder joint: Two sets of 15 repetitions of each exercise .
  * Postural correction exercises: 3 sets of postural correction were performed with 3-5 repetitions per set.
  * Scapular strengthening exercises : two sets of ten repetitions
  * The Intervention protocol: 45 to 50 minutes sessions 3 days per week for 8 week
  Arms: intercostal mulligan moblization
Other: Exercise — 1.3.b. Therapeutic Exercise:
  * Therapeutic exercise included: (prior to 3 month post mastectomy).
  * Assistive range of motion exercises (AAROME): Two sets of 15 repetitions of each exercise were performed for AAROME .
  * Active stretching: Two sets of 10 repetitions with 15- sec hold and relax times were performed for active stretching. .
  * Strengthening exercises for the shoulder joint: Two sets of 15 repetitions of each exercise .
  * Postural correction exercises: 3 sets of postural correction were performed with 3-5 repetitions per set. .
  * Scapular strengthening exercises : Strengthening exercises performed using weights were initiated with two sets of ten repetitions, beginning with a weight of 0.5kg and progressed to 0.75 and then 1 kg.
  * The Intervention protocol: 45 to 50 minutes sessions 3 days per week for 8 week

SUMMARY:
the study is to evaluate the therapeutic efficacy of intercostal mulligan Mobilization in decreasing pain and improve ROM for shoulder dysfunction Patients post mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients post modified radical mastectomy at least 3 months prior and had a limited ROM in abduction.
* Patients post mastectomy with lateral chest wall pain.
* Age ranges between 40-60 years.
* All patients had informed written consent

Exclusion Criteria:

* Receiving any previous rehabilitation programs for the upper extremities
* The presence of any type of metastases
* The presence of lymphedema
* Bilateral breast cancer surgery
* Locoregional recurrence
* Withdrawal of the consent at any time during the study for any reason

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-16 (Estimated); Primary Completion 2026-09-16 (Estimated); Study Completion 2026-09-16 (Estimated)

PRIMARY OUTCOMES:
range of motion of shoulder abducation Universal goniometer. | Universal goniometer: maximum pain free shoulder abduction was investigated in an upright position .Normal range of active movement of the shoulder 180 degree Were recorded at baseline and at the end of 8 weeks of treatment.

SECONDARY OUTCOMES:
1.4.a. Measuring shoulder function The Arabic version of DASH questionnaire | The DASH was adapted into Arabic . contains 30 items , each item has five response choices that range from 1, ''without any difficulty or no symptoms exist'' to 5, ''.Were recorded at baseline and at the end of 8 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Aya M Submitted In Partial Fulfilment of The Requirements For Master, B.Sc. of physical therapy, Principal Investigator — Cairo universty
Locations (1):
- Cario U, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salati SA, Alsulaim L, Alharbi MH, Alharbi NH, Alsenaid TM, Alaodah SA, Alsuhaibani AS, Albaqami KA. Postmastectomy Pain Syndrome: A Narrative Review. Cureus. 2023 Oct 20;15(10):e47384. doi: 10.7759/cureus.47384. eCollection 2023 Oct. PMID 38021812
- [Background] Min J, Yeon S, Ryu J, Kim JY, Yang EJ, Il Kim S, Park S, Jeon JY. Shoulder function and health outcomes in newly diagnosed breast cancer patients receiving surgery: a prospective study. Clin Breast Cancer. 2023 Jun;23(4):e247-e258. doi: 10.1016/j.clbc.2023.03.001. Epub 2023 Mar 6. PMID 36990840